CLINICAL TRIAL: NCT06978907
Title: Evaluation of the Efficacy and Safety of Lactobacillus Crispatus M247 (Crispact®) in Combination With Vaginal Laser Therapy for Improving Vaginal Microbiota Composition and Symptomatology in Menopausal Women With Atrophic Vulvovaginitis: A Prospective, Multicenter, Randomized, Controlled Clinical Trial
Brief Title: Evaluation of the Efficacy and Safety of Lactobacillus Crispatus M247 (Crispact®) With Vaginal Laser Therapy in Menopausal Women With Atrophic Vulvovaginitis (VVA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L. crispatus M247/25.04.2025
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Atrophic Vulvovaginitis
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two groups in a 2:1 (Laser-only : Laser + Crispact) Group 1: Vaginal laser therapy only. Group 2: Vaginal laser therapy + Lactobacillus crispatus M247 (Crispact®) probiotic.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal Laser Therapy Only (Active Comparator): Participants in this arm will receive three sessions of vaginal laser therapy (Monnalisa Touch® laser), administered once every 30 days.
  Interventions: Device: Monnalisa Touch® Laser Therapy
- Vaginal Laser Therapy + Lactobacillus crispatus M247 Probiotic (Experimental): Participants in this arm will receive three sessions of vaginal laser therapy (Monnalisa Touch® laser), administered once every 30 days, in combination with daily administration of Lactobacillus crispatus M247 probiotic (Crispact®) containing 20 billion CFU, taken orally once daily for three months.
  Interventions: Device: Monnalisa Touch® Laser Therapy; Combination Product: Monnalisa Touch® Laser Therapy + Lactobacillus crispatus M247 (Crispact®)

INTERVENTIONS:
Device: Monnalisa Touch® Laser Therapy — Monnalisa Touch® laser therapy is a non-ablative fractional CO2 laser applied to the vaginal mucosa to promote tissue regeneration and maintain vaginal health. Participants in this group will receive three sessions of laser therapy, one session every 30 days.
  Other Names: Vaginal Laser Therapy
Combination Product: Monnalisa Touch® Laser Therapy + Lactobacillus crispatus M247 (Crispact®) — Participants in this group will receive three sessions of Monnalisa Touch® laser therapy, one session every 30 days, along with daily administration of Lactobacillus crispatus M247 (Crispact®), a probiotic containing 20 billion CFU, taken orally for three months.
  Other Names: Laser + Probiotic Therapy
  Arms: Vaginal Laser Therapy + Lactobacillus crispatus M247 Probiotic

SUMMARY:
This randomized, controlled, prospective, multicenter study aims to evaluate the efficacy and safety of Lactobacillus crispatus M247 in combination with vaginal laser therapy for improving vaginal microbiota composition and reducing genitourinary symptoms in menopausal women with atrophic vulvovaginitis (VVA). Participants will be randomized into two groups: one receiving laser therapy alone and the other receiving laser therapy combined with daily administration of the probiotic Lactobacillus crispatus M247 (Crispact®). Primary outcomes include changes in genitourinary symptoms assessed using a validated vulvovaginal symptom questionnaire and evaluation of safety. Secondary outcomes include changes in vaginal microbiota composition.

DETAILED DESCRIPTION:
Atrophic vulvovaginitis (VVA) is a common condition affecting menopausal women, characterized by symptoms such as vaginal dryness, dyspareunia, itching, and recurrent urinary tract infections. These symptoms result from decreased estrogen levels leading to an imbalance in vaginal microbiota. Standard treatments for VVA include hormonal therapy, but this approach is often associated with adverse effects and contraindications.

This study investigates a non-hormonal approach using Lactobacillus crispatus M247 (Crispact®), a probiotic strain known for its ability to maintain a healthy vaginal microbiota, in combination with vaginal laser therapy. The study will include 75 menopausal women diagnosed with VVA who will be randomized in a 2:1 ratio, with a greater proportion allocated to the laser-only group and the remaining participants receiving laser therapy combined with the probiotic.

Primary outcomes will include changes in genitourinary symptoms assessed using a validated vulvovaginal symptom questionnaire and evaluation of safety over the study period. Secondary outcomes will include changes in vaginal microbiota composition, including Lactobacillus crispatus levels, assessed at baseline (T0) and three months (T3).

The study is approved by the Ethics Committee for Human Experimentation (CESU), University of Urbino Carlo Bo, under protocol 124_6March2025_Lactobacillus crispatus M247_Sisti, on 29.04.2025.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal women with no menstrual cycle for >12 months.
* Diagnosed with atrophic vulvovaginitis (VVA) and experiencing related symptoms (vaginal dryness, introital and profound dyspareunia, itching, burning, bleeding during intercourse).
* Symptoms related to genitourinary syndrome of menopause (GSM), including urinary urgency, increased frequency, nocturia, recurrent cystitis, or post-coital cystitis.
* Prior negative PAP test performed within one year of enrollment.
* Women who are unresponsive to or dissatisfied with prior topical estrogen therapy or who have contraindications to local and/or systemic estrogen prescription.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Presence of preneoplastic or neoplastic lesions of the cervix, vagina, or vulva.
* Active genital and/or urinary tract infections.
* Dermatological contraindications to laser therapy.
* Ongoing systemic or local hormone therapy.
* Neurological or psychiatric disorders.
* Chronic systemic diseases of autoimmune or dysmetabolic nature.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — (This study is for biological females only, not based on gender identity).
Enrollment: 75 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Change in Genitourinary Symptoms | Baseline (T0) to Month 3 (M3).
  Assessment using the Vulvovaginal Atrophy Symptom Questionnaire (VASQ), evaluating symptom severity (e.g., vaginal dryness, itching, dyspareunia, urinary symptoms) from baseline (T0) to Month 3 (M3).
Safety Assessment | Baseline (T0) to Month 3 (M3).
  Evaluation of safety and tolerability of Lactobacillus crispatus M247 based on the incidence of adverse events throughout the study period (Baseline to Month 3).

SECONDARY OUTCOMES:
Change in Vaginal Microbiota Composition (Lactobacillus crispatus Abundance) | Baseline (T0) and 3 months (T3).
  Assessment of the change in the abundance of Lactobacillus crispatus in the vaginal microbiota, measured using vaginal swab samples analyzed at baseline (T0) and after 3 months (T3).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Villa Margherita Clinic, Roma
  - Hospital State of Republic of San Marino, San Mariano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aldunate M, Srbinovski D, Hearps AC, Latham CF, Ramsland PA, Gugasyan R, Cone RA, Tachedjian G. Antimicrobial and immune modulatory effects of lactic acid and short chain fatty acids produced by vaginal microbiota associated with eubiosis and bacterial vaginosis. Front Physiol. 2015 Jun 2;6:164. doi: 10.3389/fphys.2015.00164. eCollection 2015. PMID 26082720
- [Background] Asgharpoor H, Hadizadeh-Talasaz F, Rahmani R, Rakhshandeh H, Rahmati Z. The Effect of Citrus Aurantium Vaginal Cream on Vaginal Atrophy in Postmenopausal Women: A Quasi-experimental Study. Int J Community Based Nurs Midwifery. 2024 Jan 1;12(1):32-43. doi: 10.30476/IJCBNM.2023.98670.2251. eCollection 2024 Jan. PMID 38328013
- [Background] De Seta F, Caruso S, Di Lorenzo G, Romano F, Mirandola M, Nappi RE. Efficacy and safety of a new vaginal gel for the treatment of symptoms associated with vulvovaginal atrophy in postmenopausal women: A double-blind randomized placebo-controlled study. Maturitas. 2021 May;147:34-40. doi: 10.1016/j.maturitas.2021.03.002. Epub 2021 Mar 4. PMID 33832645
- [Background] Lubian-Lopez DM, Butron-Hinojo CA, Menjon-Beltran S, Gonzalez-Mesa E, Tapiador-Albertos S, Rodriguez-Jimenez B, Fiol-Ruiz G. Effects of Non-Ablative Solid-State Vaginal Laser (SSVL) for the Treatment of Vulvovaginal Atrophy in Breast Cancer Survivors after Adjuvant Aromatase Inhibitor Therapy: Preliminary Results. J Clin Med. 2023 Aug 31;12(17):5669. doi: 10.3390/jcm12175669. PMID 37685736
- [Background] Mitchell CM, Srinivasan S, Plantinga A, Wu MC, Reed SD, Guthrie KA, LaCroix AZ, Fiedler T, Munch M, Liu C, Hoffman NG, Blair IA, Newton K, Freeman EW, Joffe H, Cohen L, Fredricks DN. Associations between improvement in genitourinary symptoms of menopause and changes in the vaginal ecosystem. Menopause. 2018 May;25(5):500-507. doi: 10.1097/GME.0000000000001037. PMID 29206774
- [Background] Muhleisen AL, Herbst-Kralovetz MM. Menopause and the vaginal microbiome. Maturitas. 2016 Sep;91:42-50. doi: 10.1016/j.maturitas.2016.05.015. Epub 2016 Jun 1. PMID 27451320